CLINICAL TRIAL: NCT03786913
Title: Quantitative Muscle Ultrasound as a Monitoring Tool of Disease Progression in Children With Inflammatory Myositis and Duchenne Muscular Dystrophy
Brief Title: Quantitative Muscle Ultrasound as a Marker of Progression in Children With Muscular Diseases
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Waleed Ahmed Salaheldeen Hassan, Assistant professor, Benha University
Other Study IDs: BenhaU122018
Record Dates: First submitted 2018-12-21; First posted 2018-12-26 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Inflammatory Myopathy; Duchenne Muscular Dystrophy
Keywords: Inflammatory myositis; Duchenne Muscular Dystrophy; Musculoskeletal ultrasound
MeSH Terms: conditions — Myositis; Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children with muscle disease: fifty children diagnosed to have inflammatory myositis or Duchenne muscular dystrophy in whom Quantitative muscle ultrasound measurements will be performed .The captured images will be analyzed for echo intensity by means of computer-assisted grayscale histogram analysis at baseline and after 24 months.
  Interventions: Diagnostic Test: Quantitative muscle ultrasound measurements
- control group: 20 healthy children matching age and sex as control group in whom Quantitative muscle ultrasound measurement will be performed at baseline
  Interventions: Diagnostic Test: Quantitative muscle ultrasound measurements

INTERVENTIONS:
Diagnostic Test: Quantitative muscle ultrasound measurements — Quantitative ultrasound measurements will be performed to biceps, forearm flexors, quadriceps and tibialis anterior according to a standard protocol; for each muscle three consecutive measurements will be made to minimize variation in echo intensity during analysis .The captured images will be analyzed offline for echo intensity by means of computer-assisted grayscale histogram analysis.

SUMMARY:
The aim of our study is to Assess skeletal muscle structural status in children with inflammatory myositis and Duchenne muscular dystrophy using musculoskeletal ultrasound and to perform a longitudinal follow up of these changes over 2 years and to assess the relation between these findings with clinical parameters, functional scales, biochemical and electromyographic tests.

DETAILED DESCRIPTION:
This study will be carried out on two groups:

• Group (I): fifty children diagnosed to have duchenne muscular dystrophy and inflammatory myositis.

Group (II): including 20 healthy children matching age and sex as control group.

patients will be subjected to

(A) Clinical evaluation

1. Complete history taking.
2. Thorough clinical examination.
3. Body mass index (BMI) assessment.
4. Quantitative muscle strength tests
5. Functional grading
6. Childhood Myositis Assessment Scale. 7 (B) Laboratory assessment:

All patients will be subjected to the following measurements:

1. Serum creatine kinase levels (CK).
2. Serum Lactate dehydrogenase levels
3. Serum of Liver enzymes (SGOT& SGPT) levels.

(C) Electromyographic (EMG) assessment:

(D) Musculoskeletal ultrasound assessment (E) Statistical analysis

ELIGIBILITY:
Inclusion Criteria:

* children with Duchenne muscular dystrophy (DMD). Diagnosis with DMD was established according to DMD diagnostic criteria (Jennekens et al., 1991).
* children with juvenile dermatomyositis (JDM) according to Bohan and Peter diagnostic criteria ( (Bohan and Peter, 1975).

Exclusion Criteria:

* Patients with age less than 2 years were excluded from the study due to inability to perform manual muscle testing and functional scales.
* If no final diagnosis could be established.
* The presence of a concomitant illness that may result in peripheral neuropathy or myopathy.

Ages: 2 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: the study will be performed on 2 groups Group (I): fifty children diagnosed to have inflammatory myositis and Duchenne muscular dystrophy Group (II): including 20 healthy children matching age and sex as control group.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2019-02-02 (Actual); Study Completion 2019-02-02 (Actual)

PRIMARY OUTCOMES:
Kendall's manual muscle testing | 24 months
  Kendall's 0 -10 point scale measures strength of each muscle group score 0 is the weakest (worst) and 10 is the strongest (best). The following muscles were tested bilaterally: the biceps brachii muscle (BB), the forearm flexors (FF), the rectus femoris muscle (RF), the tibialis anterior muscle (TA)
Childhood myositis assessment scale | 24 months
  used to assess the severity of muscle involvement in children with dermatomyositis. The scores for the 14 items are summated to give a total score ranging from 0 (worst) to 52 (best)
Serum creatine kinase (CK) levels | 24 months
  CK measured in U/L using ELISA
Serum Lactate dehydrogenase (LDH) levels | 24 months
  CK measured in IU/L using ELISA
Aspartate aminotransferase (AST) | 24 MONTHS
  AST measured in U/L using ELISA
alanine aminotransferase (ALT) | 24 months
  ALT measured in U/L using ELISA
motor unit potential (MUP) duration | 24 months
  quantitative electromyography (QEMG) in the most affected rectus femoris and biceps brachii muscles will be performed and The motor unit potentials will be reviewed offline for the needle-detected EMG signals will be analyzed by the device software for the MUP duration measured in milliseconds.
motor unit peak-to-peak amplitude | 24 months
  quantitative electromyography (QEMG) in the most affected rectus femoris and biceps brachii muscles will be performed and The motor unit potentials will be reviewed offline for the needle-detected EMG signals will be analyzed by the device software for the peak-to-peak amplitude measured in microvolt
motor unit area to amplitude ratio (AAR) | 24 months
  quantitative electromyography (QEMG) in the most affected rectus femoris and biceps brachii muscles will be performed and The motor unit potentials will be reviewed offline for the needle-detected EMG signals will be analyzed by the device software for the motor unit AAR .

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Hassan, MD, Principal Investigator — Benha university- Qaluibya- Egypt
Locations (1):
- Benha University Hospital, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No